CLINICAL TRIAL: NCT06244537
Title: Study on the Safety and Efficacy of MR-Linac Technique in Patients With Unresectable Locally Advanced Colon Cancer
Acronym: UNLACC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Qian Peng, chief physician, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCHEC-02-2024-017
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Safety and Efficacy
Keywords: MR-Linac; unresectable locally advanced colorectal cancer; neoadjuvant radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-linac (Experimental): Patients enrolled will be treated with MR-Linac with short course radiotherapy (25Gy/5F), followed by 4 cycles of mFOLFOX6 or 3 cycles of XELOX chemotherapy, then radical surgical resection, and then postoperatively with 8 cycles of mFOLFOX6 or 5 cycles of XELOX chemotherapy.
  Interventions: Radiation: MR-linac

INTERVENTIONS:
Radiation: MR-linac — Patients enrolled will be treated with MR-Linac with short course radiotherapy (25Gy/5F), followed by 4 cycles of mFOLFOX6 or 3 cycles of XELOX chemotherapy, then radical surgical resection, and then postoperatively with 8 cycles of mFOLFOX6 or 5 cycles of XELOX chemotherapy.

SUMMARY:
In this phase I single-arm clinical study, 20 patients with T4 unresectable locally advanced colon cancer are proposed to be enrolled, who will be treated with MR-Linac with short course radiotherapy (25Gy/5F), followed by 4 cycles of mFOLFOX6 or 3 cycles of XELOX chemotherapy, then radical surgical resection, and then postoperatively with 8 cycles of mFOLFOX6 or 5 cycles of XELOX. The study will assess patients' surgical R0 resection rate, pCR or cCR rate, PFS, OS, and related adverse effects of treatment, aiming to explore the feasibility, safety, and efficacy of MR-Linac in the treatment of unresectable locally advanced colon cancer.

DETAILED DESCRIPTION:
Pre-specified run-in/feasibility phase. As outlined in the registered protocol, this record includes an initial feasibility (run-in) phase conducted under the same eligibility criteria and intervention as the definitive efficacy/safety phase. The run-in is designed solely to evaluate operational and workflow feasibility. The run-in is not powered for efficacy and will not test efficacy or survival hypotheses.

Pre-specified feasibility thresholds for proceeding include, for example: protocol adherence ≥85-90%, adaptive-plan success ≥80-90%, and accrual feasibility ≥80% of the target. The run-in sample size is capped (≈24 patients), and its endpoints/time frames are listed under Outcome Measures. Meeting these thresholds triggers continuation to the definitive phase without changing the intervention or eligibility.

ELIGIBILITY:
Inclusion criteria:

1. Patients over 18 years old
2. Patients can remain in a stationary position on the treatment bed for 1-1.5 hours
3. ECOG score 0-1
4. Pathological diagnosis of colon adenocarcinoma, clinical stage cT4N0-2M0
5. Organ function is normal, and the following conditions are required: white blood cell count ≥3.5×10^9/L; platelet count ≥100×10^9/L; hemoglobin ≥90g/L. Total bilirubin level ≤1.5× upper limit of normal (ULN); AST and ALT levels ≤2.5 × ULN; endogenous creatinine clearance rate: 56-122ml/min; serum creatinine <1.0× ULN; serum albumin ≥30g/L.
6. Able to adhere to the study protocol during the research period
7. Signed written informed consent

Exclusion Criteria:

1. Patients with dMMR or MSI-H
2. Presence of other types of tumors in addition to colon adenocarcinoma
3. Claustrophobia or inability to undergo MRI or treatment due to the presence of metal implants or other reasons
4. Distant metastasis (M1)
5. Pregnant or lactating women
6. Previous anti-tumor treatment
7. Concurrent use of prohibited drugs for treatment
8. Known history of positive human immunodeficiency virus testing or known acquired immunodeficiency syndrome.
9. Clinically significant (i.e., active) cardiovascular disease: cerebrovascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina pectoris, congestive heart failure (≥New York Heart Association class II) or severe arrhythmia requiring medication treatment
10. Individuals with uncontrolled epilepsy, central nervous system disorders or a history of mental illness, whose clinical severity may hinder signing informed consent or affect patient compliance with oral medication according to the investigator's judgement
11. Organ transplant surgery requiring immunosuppressive therapy
12. Severe, uncontrolled recurrent infections or other severe, uncontrolled comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI-linac Treatment Completion Rate | 2 years
  Is adaptive radiotherapy guided by MRI feasible for patients with locally advanced unresectable colon cancer. The feasibility of each patient will be recorded as a binary variable (1=feasible; 0=not feasible). Completion Rate = Number of Completions / Total ITT Enrollment
Clinical complete response (cCR) | 2 years
  Clinical complete response refers to the absence of detectable tumor clinically after treatment. Number of cCR cases/Number of cases completed for follow-up evaluation
Pathological complete response (pCR) | 2 years
  Pathological complete response is defined as the absence of any signs of cancer in tissue samples after treatment. Number of pCR cases / Number of completed surgeries

SECONDARY OUTCOMES:
Toxicity reaction (CTC 4.0 standard） | long range
  CTC 4.0, also known as Common Terminology Criteria for Adverse Events version 4.0, is an extensively used classification system for assessing drug toxicity. This system categorizes drug toxicity into five levels: Grade 0, Grade 1, Grade 2, Grade 3, and Grade 4.
R0 resection rate | 2 years
  During surgery, the R0 resection rate refers to the complete removal of the entire tumor with no residual abnormalities present in the surrounding normal tissue. R0 rate = Number of R0 cases / Total number of surgical procedures performed
Surgical complications | 2 years
  Surgical complications refers to adverse events or problems that arise during or after a surgical procedure. These complications can range from minor issues to serious complications that may have significant consequences for the patient.
Local control rate | 2 years
  Proportion of cases in remission and stable disease after treatment, i.e., proportion of patients who did not experience disease progression.
Disease-free survival | 2 years
  The time from the start of treatment to the first tumor recurrence/metastasis, or death of the subject due to any cause.
Overall survival | 2 years
  Time from the start of the patient's treatment to the patient's death from any cause

OTHER OUTCOMES:
Online adaptation time, compliance rate, technical success rate | 8 months.
  This pilot analysis was pre-specified in the registered protocol as an initial feasibility/run-in phase. Number of successful cases with the initial feasibility/run-in phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital & Institute, Affiliated Cancer Hospital of University of Electronic Science and Technology of China., Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Cao W, Chen HD, Yu YW, Li N, Chen WQ. Changing profiles of cancer burden worldwide and in China: a secondary analysis of the global cancer statistics 2020. Chin Med J (Engl). 2021 Mar 17;134(7):783-791. doi: 10.1097/CM9.0000000000001474. PMID 33734139
- [Background] Yoshihara M, Hiyama T, Tanaka S. [Epidemiology of colorectal cancer]. Nihon Naika Gakkai Zasshi. 2007 Feb 10;96(2):200-6. doi: 10.2169/naika.96.200. No abstract available. Japanese. PMID 17370582
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Schmoll HJ, Van Cutsem E, Stein A, Valentini V, Glimelius B, Haustermans K, Nordlinger B, van de Velde CJ, Balmana J, Regula J, Nagtegaal ID, Beets-Tan RG, Arnold D, Ciardiello F, Hoff P, Kerr D, Kohne CH, Labianca R, Price T, Scheithauer W, Sobrero A, Tabernero J, Aderka D, Barroso S, Bodoky G, Douillard JY, El Ghazaly H, Gallardo J, Garin A, Glynne-Jones R, Jordan K, Meshcheryakov A, Papamichail D, Pfeiffer P, Souglakos I, Turhal S, Cervantes A. ESMO Consensus Guidelines for management of patients with colon and rectal cancer. a personalized approach to clinical decision making. Ann Oncol. 2012 Oct;23(10):2479-2516. doi: 10.1093/annonc/mds236. PMID 23012255
- [Background] Wu C. Systemic Therapy for Colon Cancer. Surg Oncol Clin N Am. 2018 Apr;27(2):235-242. doi: 10.1016/j.soc.2017.11.001. Epub 2017 Dec 16. PMID 29496087
- [Background] Karoui M, Rullier A, Luciani A, Bonnetain F, Auriault ML, Sarran A, Monges G, Trillaud H, Le Malicot K, Leroy K, Sobhani I, Bardier A, Moreau M, Brindel I, Seitz JF, Taieb J. Neoadjuvant FOLFOX 4 versus FOLFOX 4 with Cetuximab versus immediate surgery for high-risk stage II and III colon cancers: a multicentre randomised controlled phase II trial--the PRODIGE 22--ECKINOXE trial. BMC Cancer. 2015 Jul 10;15:511. doi: 10.1186/s12885-015-1507-3. PMID 26156156
- [Background] Chang H, Yu X, Xiao WW, Wang QX, Zhou WH, Zeng ZF, Ding PR, Li LR, Gao YH. Neoadjuvant chemoradiotherapy followed by surgery in patients with unresectable locally advanced colon cancer: a prospective observational study. Onco Targets Ther. 2018 Jan 17;11:409-418. doi: 10.2147/OTT.S150367. eCollection 2018. PMID 29398921
- [Background] Tomizawa K, Miura Y, Fukui Y, Hanaoka Y, Toda S, Moriyama J, Inoshita N, Ozaki Y, Takano T, Matoba S, Kuroyanagi H. Curative resection for locally advanced sigmoid colon cancer using neoadjuvant chemotherapy with FOLFOX plus panitumumab: A case report. Int J Surg Case Rep. 2017;31:128-131. doi: 10.1016/j.ijscr.2017.01.027. Epub 2017 Jan 17. PMID 28135678
- [Background] Reima H, Soplepmann J, Elme A, Lohmus M, Tiigi R, Uksov D, Innos K. Changes in the quality of care of colorectal cancer in Estonia: a population-based high-resolution study. BMJ Open. 2020 Oct 8;10(10):e035556. doi: 10.1136/bmjopen-2019-035556. PMID 33033081
- [Background] Foxtrot Collaborative Group. Feasibility of preoperative chemotherapy for locally advanced, operable colon cancer: the pilot phase of a randomised controlled trial. Lancet Oncol. 2012 Nov;13(11):1152-60. doi: 10.1016/S1470-2045(12)70348-0. Epub 2012 Sep 25. PMID 23017669
- [Background] Reibetanz J, Germer CT. [Neoadjuvant chemotherapy for locally advanced colon cancer : Initial results of the FOxTROT study.]. Chirurg. 2013 Oct 13. doi: 10.1007/s00104-013-2631-8. Online ahead of print. No abstract available. German. PMID 24122133
- [Background] Karoui M, Rullier A, Piessen G, Legoux JL, Barbier E, De Chaisemartin C, Lecaille C, Bouche O, Ammarguellat H, Brunetti F, Prudhomme M, Regimbeau JM, Glehen O, Lievre A, Portier G, Hartwig J, Goujon G, Romain B, Lepage C, Taieb J; for PRODIGE 22 investigators/collaborators. Perioperative FOLFOX 4 Versus FOLFOX 4 Plus Cetuximab Versus Immediate Surgery for High-Risk Stage II and III Colon Cancers: A Phase II Multicenter Randomized Controlled Trial (PRODIGE 22). Ann Surg. 2020 Apr;271(4):637-645. doi: 10.1097/SLA.0000000000003454. PMID 31356278
- [Background] Ryan R, Gibbons D, Hyland JM, Treanor D, White A, Mulcahy HE, O'Donoghue DP, Moriarty M, Fennelly D, Sheahan K. Pathological response following long-course neoadjuvant chemoradiotherapy for locally advanced rectal cancer. Histopathology. 2005 Aug;47(2):141-6. doi: 10.1111/j.1365-2559.2005.02176.x. PMID 16045774
- [Background] Huang CM, Huang MY, Ma CJ, Yeh Y-, Tsai HL, Huang CW, Huang CJ, Wang JY. Neoadjuvant FOLFOX chemotherapy combined with radiotherapy followed by radical resection in patients with locally advanced colon cancer. Radiat Oncol. 2017 Mar 7;12(1):48. doi: 10.1186/s13014-017-0790-3. PMID 28270172
- [Background] Venigalla S, Chowdhry AK, Wojcieszynski AP, Lukens JN, Plastaras JP, Metz JM, Ben-Josef E, Mahmoud NN, Reiss KA, Shabason JE. Comparative Effectiveness of Neoadjuvant Chemoradiation Versus Upfront Surgery in the Management of Recto-Sigmoid Junction Cancer. Clin Colorectal Cancer. 2018 Sep;17(3):e557-e568. doi: 10.1016/j.clcc.2018.05.005. Epub 2018 May 17. PMID 29910004
- [Background] Krishnamurty DM, Hawkins AT, Wells KO, Mutch MG, Silviera ML, Glasgow SC, Hunt SR, Dharmarajan S. Neoadjuvant Radiation Therapy in Locally Advanced Colon Cancer: a Cohort Analysis. J Gastrointest Surg. 2018 May;22(5):906-912. doi: 10.1007/s11605-018-3676-2. Epub 2018 Feb 9. PMID 29427227
- [Background] Qiu B, Ding PR, Cai L, Xiao WW, Zeng ZF, Chen G, Lu ZH, Li LR, Wu XJ, Mirimanoff RO, Pan ZZ, Xu RH, Gao YH. Outcomes of preoperative chemoradiotherapy followed by surgery in patients with unresectable locally advanced sigmoid colon cancer. Chin J Cancer. 2016 Jul 7;35(1):65. doi: 10.1186/s40880-016-0126-y. PMID 27389519
- [Background] Boldrini L, Intven M, Bassetti M, Valentini V, Gani C. MR-Guided Radiotherapy for Rectal Cancer: Current Perspective on Organ Preservation. Front Oncol. 2021 Mar 30;11:619852. doi: 10.3389/fonc.2021.619852. eCollection 2021. PMID 33859937
- [Background] Chiloiro G, Boldrini L, Meldolesi E, Re A, Cellini F, Cusumano D, Corvari B, Mantini G, Balducci M, Valentini V, Gambacorta MA. MR-guided radiotherapy in rectal cancer: First clinical experience of an innovative technology. Clin Transl Radiat Oncol. 2019 Apr 12;18:80-86. doi: 10.1016/j.ctro.2019.04.006. eCollection 2019 Sep. PMID 31341981
- [Background] Slotman B, Gani C. Online MR-guided radiotherapy - A new era in radiotherapy. Clin Transl Radiat Oncol. 2019 Apr 17;18:102-103. doi: 10.1016/j.ctro.2019.04.011. eCollection 2019 Sep. No abstract available. PMID 31341984
- [Background] Winkel D, Bol GH, Kroon PS, van Asselen B, Hackett SS, Werensteijn-Honingh AM, Intven MPW, Eppinga WSC, Tijssen RHN, Kerkmeijer LGW, de Boer HCJ, Mook S, Meijer GJ, Hes J, Willemsen-Bosman M, de Groot-van Breugel EN, Jurgenliemk-Schulz IM, Raaymakers BW. Adaptive radiotherapy: The Elekta Unity MR-linac concept. Clin Transl Radiat Oncol. 2019 Apr 2;18:54-59. doi: 10.1016/j.ctro.2019.04.001. eCollection 2019 Sep. PMID 31341976
- [Background] van Rossum PS, van Lier AL, van Vulpen M, Reerink O, Lagendijk JJ, Lin SH, van Hillegersberg R, Ruurda JP, Meijer GJ, Lips IM. Diffusion-weighted magnetic resonance imaging for the prediction of pathologic response to neoadjuvant chemoradiotherapy in esophageal cancer. Radiother Oncol. 2015 May;115(2):163-70. doi: 10.1016/j.radonc.2015.04.027. Epub 2015 May 19. PMID 26002307
- [Background] Kontaxis C, Bol GH, Kerkmeijer LGW, Lagendijk JJW, Raaymakers BW. Fast online replanning for interfraction rotation correction in prostate radiotherapy. Med Phys. 2017 Oct;44(10):5034-5042. doi: 10.1002/mp.12467. Epub 2017 Aug 9. PMID 28703497
- [Background] Intven MPW, de Mol van Otterloo SR, Mook S, Doornaert PAH, de Groot-van Breugel EN, Sikkes GG, Willemsen-Bosman ME, van Zijp HM, Tijssen RHN. Online adaptive MR-guided radiotherapy for rectal cancer; feasibility of the workflow on a 1.5T MR-linac: clinical implementation and initial experience. Radiother Oncol. 2021 Jan;154:172-178. doi: 10.1016/j.radonc.2020.09.024. Epub 2020 Sep 22. PMID 32976875